CLINICAL TRIAL: NCT04530058
Title: The Effects of Metformin on Morbidity and Mortality in Elderly Patients- a Prospective Randomized Control Trial (RCT)
Brief Title: The Effects of Metformin on Morbidity and Mortality in Elderly Patients
Acronym: MET-ELD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15230
Record Dates: First submitted 2020-07-28; First posted 2020-08-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Placebos
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg twice a day, administered orally or via gastric tube.
  Arms: Metformin
Drug: Placebos — Placebo twice a day, administered orally or via gastric tube.
  Arms: Control

SUMMARY:
Elderly patients have an increased susceptibility to burns and a substantial mortality that has not significantly changed over the last three decades. Elderly burn patients not only have an augmented response to burn but also express a prolonged hypermetabolic response.Glucose metabolism with insulin resistance is a hypermetabolic response pathway that profoundly affects post-burn outcomes. The aim if this study is to determine whether metformin can improve morbidity and mortality in elderly burn patients. The investigators hypothesize that metformin will improve clinical outcomes and mortality of elderly burn patients by alleviating the complex inflammatory and hypermetabolic responses after burn.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 - 99 years of age.
2. ≥5% total body surface area (TBSA) burn.
3. Admitted to burn center ≤ 120 hours post-burn injury.
4. At least one surgical intervention likely required.
5. Provide written informed consent.

Exclusion Criteria:

1. Death upon admission.
2. Decision not to treat due to burn injury severity.
3. Presence of anoxic brain injury that is not expected to result in complete recovery.
4. Pre-existing renal failure (eGFR is < 30 mL/min).
5. Severe liver disease (Child-Pugh C).
6. Pre-existing insulin-dependent type II diabetes.
7. Clinical contraindication to give metformin.
8. Allergy to metformin or insulin.
9. History of lactic acidosis while receiving metformin treatment.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Record mortality | Acute hospitalization up to one year post burn.
  Patient mortality will be recorded during hospitalization and outpatient follow-ups.
Record the episodes of sepsis. | daily until discharge (1-4 months post admission depending on severity of injury)]
  Patients will be assessed daily for episodes of sepsis. The total number of episodes over the course of hospital stay will be recorded.
Record episodes of infection. | daily until discharge (1-4 months post admission depending on severity of injury)]
  Patients will be assessed daily for episodes of infection. The total number of episodes over the course of hospital stay will be recorded.
Record episodes of pneumonia. | daily until discharge (1-4 months post admission depending on severity of injury)]
  Patients will be assessed daily for episodes of infection. The total number of episodes over the course of hospital stay will be recorded.
Organ function - Alkaline phosphatase (ALP) | twice weekly until discharge (1-4 months post admission depending on severity of injury)]
  Organ function will be assessed by measuring the biomarker: ALP (U/L).
Organ function - Alanine transaminase (ALT) | twice weekly until discharge (1-4 months post admission depending on severity of injury)]
  Organ function will be assessed by measuring the biomarker: ALT (U/L).
Organ function - Bilirubin | twice weekly until discharge (1-4 months post admission depending on severity of injury)]
  Organ function will be assessed by measuring the biomarker: bilirubin (umol).
Organ function - Blood Urea Nitrogen (BUN) | twice weekly until discharge (1-4 months post admission depending on severity of injury)]
  Organ function will be assessed by measuring the biomarker: BUN (mmol).
Organ function - Creatinine | twice weekly until discharge (1-4 months post admission depending on severity of injury)]
  Organ function will be assessed by measuring the biomarker: creatinine (umol/L).

SECONDARY OUTCOMES:
Measures of steady-state resting energy expenditure (REE) | weekly until discharge if a patient is intubated and ventilated (1-4 months post admission depending on severity of injury)]
  Metabolic response to injury and illness can be studied by measuring steady-state resting energy expenditure. Hypermetabolism is used as a secondary endpoint as stress-induced diabetes is associated with inflammation and hypermetabolism.
Perform oral glucose tolerance test | once at discharge from hospital (1-4 months post admission depending on the severity of injury)]
  Standard fasting oral glucose tolerance test with an intake of 75 g of glucose. Subsequent measurements (in mg/dl) of glucose in blood, insulin and c-peptide will be conducted over 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Jeschke, MD PhD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No